CLINICAL TRIAL: NCT02659280
Title: Using "Store and Forward" Tele-health as an Adjunct to Traditional Outpatient or Home Health Physical Therapy
Acronym: TELE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: Hennepin County Medical Center, Minneapolis (Other); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MinneapolisMRF
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Chronic Disease
Keywords: telerehabilitation
MeSH Terms: conditions — Chronic Disease | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care Therapy (Active Comparator): Home Health or Outpatient Physical therapy services (a minimum of 1x/week).
  Interventions: Other: Standard of Care
- Adjunct Therapy (Experimental): Home Health or Outpatient Physical therapy services (a minimum of 1x/week) with an adjunct Home Exercise Program given up to 1x/wk via "Store and Forward" tele-health through the Hudl Technique app.
  Interventions: Other: Adjunct Therapy

INTERVENTIONS:
Other: Adjunct Therapy — "Store and Forward" Tele-heath
  Arms: Adjunct Therapy
Other: Standard of Care — Standard of Care Outpatient Physical Therapy
  Arms: Standard of Care Therapy

SUMMARY:
This study will take about 3-16 months. Participants will be inpatients in the Hennepin Health System that are transitioning into outpatient or home health Physical Therapy or current outpatient patients. Investigators will assess 24 participants for eligibility based on the study's inclusion criteria. If eligible, Investigators will attain informed consent and provide instruction on how to use a coaching app, Hudl Technique, and enter data in the Apple Health Kit (all participants will be gifted an iPad mini 4, cover and Hudl Technique app). Baseline Body Mass Index (BMI) will be taken and entered in the Apple Health Kit. Randomization (1:1) will occur by an outside statistician. 12 patients will be allotted to the control group (receive traditional Outpatient PT and have access to the Apple Health Kit and Hudl Technique with the gifted iPad). 12 patients will be the variable group (receive traditional Outpatient PT, have access to the Apple Health Kit and Hudl Technique with the gifted iPad, and have an adjunct Home Exercise Program which will be administered via tele-health "store and forward" technology 1x/wk). There will be an 8 week assessment in which investigators plan to measure 1) satisfaction with PT (via survey) 2) Home Exercise Program (HEP) compliance (via survey) 3) incidents of ED visits or hospital admissions 4) BMI (via patient report with option to put it in the Apple Health Kit). There will be a 24 week assessment in which investigators will measure the same 4 measurements. Investigators plan on performing this protocol for an additional 24 participants in late 2016/early 2017 (48 participants in total). Unfortunately, this will be a non-blinded (assessor, therapist and participant) study due to the nature of the intervention and how investigators received the funding. Casey Byron will be the Principal Investigator. Investigators would like the statistician to be blinded to group allocation until completion of the study (roughly 3/11/2017).

DETAILED DESCRIPTION:
Hennepin Health System (HHS) will determine participant's eligibility in the pilot project if a participant meets the following stipulations; 1) The prospective participant must be an Hennepin Health Services outpatient or home health Physical Therapy (PT) patient. 2) The prospective participant's primary PT and Primary Investigator must determine that the participant has adequate motor control to participate in a HEP (home exercise program) on their own. 3) The prospective participant's primary PT and Primary Investigator must determine that the prospective participant has adequate cognitive ability to use electronic assistive technology (iPad Mini 4). The prospective participant will need to live greater than 100 miles from Minneapolis and/or needs to have financial hardship (as designated by being on Medical Assistance, Emergency Medical Assistance, Hennepin Care, Medicaid, Medical Assistance Cost Plan, Wavered services or have no health insurance).

Note: The prospective participant may receive home health or outpatient PT at another facility other than Hennepin Health System (HHS), if they are from greater than 100 miles from Minneapolis (but the participant's care will need to be tied to a HHS admission).

The tele-health will be administered in the following manner;

1. The participant's primary PT will determine the appropriateness for this adjunct therapy and contact the tele-therapist/Primary Investigator, Casey Byron, MPT.
2. Casey Byron, MPT will perform a chart review and interview the participant to determine if they meet eligibility requirements.
3. Participant will sign the pilot program contract agreement, informed consent agreement and terms and conditions for the Hudl Technique app. The participant will be given information on how to operate the iPad Mini 4, how to use the Hudl Technique app and be given information on what to do if problems occur.
4. The participant's primary PT will discuss the home exercise program (HEP) that they wish for the participant to perform with the tele-therapist.
5. The tele-therapist will formulate an audio/video clip through Hudl Technique of the HEP and send it to the participant.
6. The participant will record their performance of the HEP using the Hudl Technique app, iPad Mini 4 and iPad Mini 4 tripod and send their audio/video clip back to the tele-therapist.
7. The video clip will be analyzed by the tele-therapist. Hudl Technique tools such as slow motion video, comparing two videos side by side, measuring angles, highlighting points of emphasis, and an audio voice over will be used to formulate a critiqued video clip.
8. The critiqued video clip will be sent back to the participant.
9. The participant will view the critiqued video clip and await the next video. ***There will be a maximum of 1 HEP per week.***
10. The tele-health PT and participant's primary PT will correspond for updates to participant's HEP.
11. The critiqued video clip will be "deleted" from the tele-therapists Hudl Technique account (HHS will not store any video clips that we generate).

Study Parameters to be Measured:

Participants will need to agree to data analytics of their electronic medical record (EMR). We will need access to information like payer source, diagnoses, address, and past and future emergency department and inpatient visits to the hospital. This will be performed through EMR review here at HHS and a survey for participants living greater than 100 miles from Minneapolis. The Hudl Technique app and a survey will allow for measurement of adherence to HEP. Participant's satisfaction with tele-health will be measured via survey (Modified Patient Satisfaction with Outpatient Physical Therapy Scale)1. Participants would be encouraged to allow the use of the Apple Health Kit. Participants would be encouraged to enter data in the Apple Health Kit, on a regular basis. This IOS/Apple program would allow for the measurement of changes that occur to a participant's body measurements (height, weight, and body mass index) with this adjunct therapy. The participant's use of the Apple Health Kit would be voluntary. Body weight measurements would also be assessed via survey.

ELIGIBILITY:
Inclusion Criteria:

* Hennepin Health System (HHS) will determine participant's eligibility in the pilot project if a participant meets the following stipulations
* The prospective participant must be an HHS outpatient or home health Physical Therapy (PT) patient.
* The prospective participant's primary PT must determine that the participant has adequate motor control to participate in a HEP (home exercise program) on their own.
* The prospective participant has adequate cognitive ability to use electronic assistive technology (iPad Mini
* The prospective participant will need to live greater than 100 miles from Minneapolis and/or needs to have financial hardship (as designated by being on Medical Assistance, Emergency Medical Assistance, Hennepin Care, Medicaid, Medical Assistance Cost Plan, Wavered services or have no health insurance).

Exclusion Criteria:

* Any participant less than the age of 18 years of age. Any participant who is pregnant or has reason to beleive they are pregnant,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Improved compliance with Physical Therapy Home Exercise Program | 24 weeks
  Subjects will have statistically significant improvement in the frequency of performing their Home Exercise Program (HEP). This will be measured via survey with the modified Patient Satisfaction for Outpatient Physical Therapy Survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beattie PF, Pinto MB, Nelson MK, Nelson R. Patient satisfaction with outpatient physical therapy: instrument validation. Phys Ther. 2002 Jun;82(6):557-65. PMID 12036397
- [Derived] Van de Winckel A, Nawshin T, Byron C. Combining a Hudl App With Telehealth to Increase Home Exercise Program Adherence in People With Chronic Diseases Experiencing Financial Distress: Randomized Controlled Trial. JMIR Form Res. 2021 Mar 18;5(3):e22659. doi: 10.2196/22659. PMID 33640865